CLINICAL TRIAL: NCT02888847
Title: Effect of High Light Intensity Bleaching Protocol Versus Descending Light Intensities Bleaching Protocol on Post Bleaching Teeth Sensitivity: A Randomized Clinical Trial
Brief Title: High Light Intensity Bleaching Versus Descending Light Intensities Bleaching on Post Bleaching Teeth Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: British University In Egypt (Other)
Responsible Party: Principal Investigator, Shadwa Hatem Saad Kabil, Shadwa Hatem Saad Kabil, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CEBD-CU-2016-08-195
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Discoloured Teeth
Keywords: post bleaching teeth sensitivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Philips Zoom! White Speed whitening lamp (Active Comparator): Philips Zoom! White Speed whitening lamp
  Interventions: Device: Philips Zoom! White Speed whitening lamp
- Philips Zoom! Advanced power lamp (Sham Comparator): Philips Zoom! Advanced power whitening lamp
  Interventions: Device: Philips Zoom! Advanced power whitening lamp

INTERVENTIONS:
Device: Philips Zoom! White Speed whitening lamp — bleaching protocol with descending built in light intensities
  Arms: Philips Zoom! White Speed whitening lamp
Device: Philips Zoom! Advanced power whitening lamp — bleaching protocol with high light intensity
  Arms: Philips Zoom! Advanced power lamp

SUMMARY:
Compare teeth sensitivity using bleaching protocol with different light intensities (Philips Zoom!™ White Speed whitening gel and lamp, Discus Dental, Inc., Culver City, CA, USA.) versus bleaching protocol with the same light intensity (Philips Zoom!™ Advanced Power whitening gel and lamp, Discus Dental, Inc., Culver City, CA, USA.).

DETAILED DESCRIPTION:
This study will be applied to patients suffering from teeth discolorations. Nowadays, vital tooth bleaching is one of the most requested cosmetic dental procedures asked by patients who want and aesthetically more pleasing smile. The American Dental Association (ADA) has advised patients to ask the dentists to adamant the most suitable bleaching treatment, especially for those complaining of tooth sensitivity, dental restorations, extremely dark discolorations, and single dark teeth.

Tooth sensitivity (TS) is the most common clinical side effect of tooth bleaching. Tooth sensitivity (TS) caused by bleaching procedures usually results in mild and transient pain; however, it can occasionally cause significant discomfort that is a main deterrent to patients successfully completing bleaching treatments. Considering that TS has been reported as a common side effect, affecting more than 60% of the patients that undergo this cosmetic treatment. Greater tooth sensitivity has been reported with in-office bleaching with adjunct light compared with no light. Existing literature reveals that activation of bleaching agents by heat or light may have an adverse effect on pulpal tissue. It was already reported that the use of intense lights does elevate bleach temperature, but it results in increased intrapulpal temperatures, which may further impact patient sensitivity and pulpal health.Hence, in this study different light intensities bleaching protocol will be used aiming at overcoming this complication.

ELIGIBILITY:
Inclusion Criteria:

1. Patients included in this clinical trial were at least18 years old.
2. Patients should be free from any systemic disease that may affect normal healing and predictable outcome.
3. Patients who will agree to the consent and will commit to follow-up period.
4. Willing to refrain from tobacco products and any colored liquids or food (e.g. coffee, tea, tomato sauce etc.) during the active study period.

Exclusion Criteria:

1. Patients with any systemic disease that may affect normal healing.
2. Patient with bad oral hygiene.
3. Pregnant females.
4. Patients who could/would not participate in a 3month follow-up.
5. Untreated periodontal disease were not allowed.
6. Active caries or defective Restorations in 6 anterior teeth.
7. Sensitive Teeth
8. Bleaching history
9. Patients participating in more than 1 dental study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-11-10 (Actual)

PRIMARY OUTCOMES:
post bleaching teeth sensitivity | after 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- British Unibersity in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided